CLINICAL TRIAL: NCT06175923
Title: Role of the BMP Pathway in Myelodysplastic Syndromes Progression and in the Transition to Acute Myeloid Leukemia
Brief Title: Role of BMP Pathway in MDS Progression
Acronym: BMP-MDS
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0491
Record Dates: First submitted 2023-11-29; First posted 2023-12-19 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-11

CONDITIONS: Myelodysplastic Syndromes; Acute Myelogenous Leukemia
Keywords: BMP; MSC; MDS; microenvironment
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone marrow aspirates will be collected, both at diagnosis and 6-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDS patients: Adult patients with myelodysplastic syndrome or suspected myelodysplastic syndrome according to the criteria defined by the World Health Organization:
  * one or more cytopenias,
  * and/or dysplasia of one or more lines,
  * and/or bone marrow blastosis
  * and/or sideroblasts in medullary crowns
  * and/or genetic/cytogenetic abnormalities characteristic of MDS.
  * Whatever the R-IPSS stage (Revised International Prognostic Scoring System)
  * No history of cytotoxic treatment (hydroxycarbamide, azacytidine)
  Interventions: Biological: Collection of EDTA (disodium salt of ethylenediaminetetraacetic acid) tubes of marrow during routine care
- AML patients: Adult patients with suspected de novo acute myeloid leukemia at initial management
  Interventions: Biological: Collection of EDTA (disodium salt of ethylenediaminetetraacetic acid) tubes of marrow during routine care

INTERVENTIONS:
Biological: Collection of EDTA (disodium salt of ethylenediaminetetraacetic acid) tubes of marrow during routine care — When bone marrow is collected as part of a patient's care (diagnosis, follow-up, suspected AML/MDS hemopathy), one or two additional EDTA tubes of marrow are collected. Certain hematological data (NFP, genetic and molecular characteristics) will be collected in anonymized form and correlated with the BMP pathway alterations measured.

SUMMARY:
Myelodysplastic syndromes (MDS) are hematological cancers that can progress to acute myelogenous leukemia (AML). The involvement of the microenvironment in the maintenance, resistance and evolution of MDS is increasingly described.

The Bone Morphogenetic Protein (BMP) pathway is involved in numerous functions, including self-renewal of the hematopoietic stem cell compartment and the regulation of hematopoiesis, via interaction with bone marrow stromal cells. Investigators have demonstrated its involvement in chronic myeloid leukemia (CML) and AML, in particular via the activation of TWIST1, ΔNp73, NANOG; it is responsible for an increased state of quiescence of certain cancer stem cells and their resistance.

Preliminary results based on the analysis of large databases suggest that the BMP pathway is also altered early in MDS. This study explores the alteration of this pathway in MDS and its involvement in the transformation into AML.

If appropriate, the BMP pathway could constitute a very promising therapeutic target to combat transformation into AML.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with myelodysplastic syndrome or suspected myelodysplastic syndrome according to the criteria defined by the World Health Organization Or
* Adult patient with suspicion of de novo acute myeloid leukemia at initial treatment

Exclusion Criteria:

* Frontier MDS/myeloproliferative syndromes including chronic myelomonocytic leukemia
* MDS and AML having already benefited from cytotoxic treatment including hydroxycarbamide, azacytidine, intensive chemotherapy
* Patients objecting to their inclusion in the study
* Pregnant or breastfeeding women
* Patients under legal protection measure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult patients with untreated myelodysplastic syndromes at risk of progression to acute myeloid leukemia.
  * Adult patients with de novo AML
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-27 (Estimated); Primary Completion 2029-01-27 (Estimated); Study Completion 2034-01-27 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of the BMP pathway : Bone marrow plasma BMP2/BMP4 levels | at diagnosis, at 6 months, at 5 years
  Descriptive analysis of the BMP pathway in bone marrow-derived cells from MDS patients at the protein, transcriptomic and functional levels :
  Marrow plasma to study the concentration of cytokines of interest BMP2 and BMP4
Descriptive analysis of the BMP pathway : Bone marrow mononuclear cell fraction | at diagnosis, at 6 months, at 5 years
  Descriptive analysis of the BMP pathway in bone marrow-derived cells from MDS patients at the protein, transcriptomic and functional levels :
  Medullary blood mononuclear cells: expression of membrane receptors BMPRIA and BMPRIB by RT-QPCR and flow cytometry, expression of cytokines BMP2 and BMP4 (RT-QPCR), degree of phosphorylation of SMAD intermediates by western blot and/or flow cytometry, expression of BMP pathway target genes by RT-QPCR
Descriptive analysis of the BMP pathway : - Bone marrow mesenchymal stem cells number and differentiation capacities after passage 0 - Functional level | at diagnosis, at 6 months, at 5 years
  Descriptive analysis of the BMP pathway in bone marrow-derived cells from MDS patients at functional level :
  Medullary MSCs will be cultured and studied from functional angle (culture, colony-forming units tests, long term culture initiating colony)
Descriptive analysis of the BMP pathway : - Bone marrow mesenchymal stem cells number and differentiation capacities after passage 0 - Transcriptomic level | at diagnosis, at 6 months, at 5 years
  Descriptive analysis of the BMP pathway in bone marrow-derived cells from MDS patients at transcriptomic level :
  Medullary MSCs will be cultured and studied from transcriptomic angle (expression of receptors, BMP cytokines, target genes, etc.).
Descriptive analysis of the BMP pathway : - Bone marrow mesenchymal stem cells number and differentiation capacities after passage 0 - Protein level | at diagnosis, at 6 months, at 5 years
  Descriptive analysis of the BMP pathway in bone marrow-derived cells from MDS patients at the protein level :
  Medullary MSCs will be cultured and studied from protein angle (cytokines present in the supernatant).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No